CLINICAL TRIAL: NCT06118034
Title: Effect of Colchicine on Perioperative Anti-inflammatory Organ Injury in Cardiac Surgery : a Multi-center, Randomized, Controlled, Double-blind Clinical Trial
Brief Title: Effect of Colchicine on Perioperative Anti-inflammatory Organ Injury in Cardiac Surgery
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Collaborators: First Affiliated Hospital of Zhejiang University (Other); Jinan Central Hospital (Other); The First People's Hospital of Changzhou (Other); Xinhua hospital of ILi in Kazakhstan automomous district (Unknown); First Affiliated Hospital of Harbin Medical University (Other); The Affiliated Hospital of Yangzhou University (Unknown); Shandong Provincial Hospital (Other Government); The First People's Hospital of Huai'an (Unknown); The First Affiliated Hospital of Shihezi University Medical College (Unknown); Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-LCYJ-ZD-03
Record Dates: First submitted 2023-10-24; First posted 2023-11-07 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Inflammatory Response; Cardiac Disease
MeSH Terms: conditions — Heart Diseases | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (colchicine group) (Experimental): The experimental group take 0.5mg of colchicine tablets orally for 3 days before surgery, and continue to take 0.5mg every other day (qod) for 10 days after tracheal extubation.
  Interventions: Drug: Colchicine 0.5 MG
- Control group (Placebo Comparator): The control group take 0.5mg of placebo tablets orally for 3 days before surgery, and continue to take 0.5mg every other day (qod) for 10 days after tracheal extubation.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine 0.5 MG — Take 0.5mg of colchicine tablets orally for 3 days before surgery, and continued to take 0.5mg every other day (qod) for 10 days after tracheal extubation.
  Other Names: Routine cardiovascular surgery and peri-operative management
  Arms: Experimental group (colchicine group)
Drug: Placebo — Take 0.5mg of starch tablets orally for 3 days before surgery, and continued to take 0.5mg every other day (qod) for 10 days after tracheal extubation.
  Other Names: Routine cardiovascular surgery and peri-operative management
  Arms: Control group

SUMMARY:
All patients will be completed collection of demographic data, clinical data, and be observed for inflammatory organ damage, oxygenation index or SpO2/ FIO2, WBC, NEU, interleukin-1β, interleukin-6, interleukin-8 (IL-1β/6/8), tumor necrosis factor-α (TNF-α), C-reactive protein (CRP), procalcitonin (PCT), myoglobin (Myo), creatine kinase-MB (CK-MB), high-sensitivity cardiac troponin T (hs-cTnT), neutrophil elastase (NE), myeloperoxidase (MPO), APACHE II score, alanine transaminase (ALT), aspartate transaminase (AST), total bilirubin, Murray lung injury score, serum creatinine, eGFR, mechanical ventilation time, ICU length of stay, drug-related gastrointestinal reactions, and 30-day and 90-day all-cause mortality, among other indicators.

DETAILED DESCRIPTION:
This study is a multicenter, randomized, controlled, double-blind, placebo- controlled clinical trial. A total of 768 patients who met the inclusion and exclusion criteria and were scheduled for cardiac surgery under cardiopulmonary bypass were enrolled. After signing informed consent, patients were randomly divided into the experimental group and the control group. Patients in the experimental group took 0.5mg of colchicine tablets orally for 3 days before surgery and continued to take 0.5mg daily for 10 days after tracheal extubation. Patients in the control group received an equivalent amount of starch placebo tablets, administered at the same times and in the same doses as the experimental group, during the colchicine/placebo treatment period, without affecting the patients' standard treatment protocols.

All patients will be completed collection of demographic data, clinical data, and be observed for inflammatory organ damage, oxygenation index or SpO2/ FIO2, WBC, NEU, interleukin-1β, interleukin-6, interleukin-8 (IL-1β/6/8), tumor necrosis factor-α (TNF-α), C-reactive protein (CRP), procalcitonin (PCT), myoglobin (Myo), creatine kinase-MB (CK-MB), high-sensitivity cardiac troponin T (hs-cTnT), neutrophil elastase (NE), myeloperoxidase (MPO), APACHE II score, alanine transaminase (ALT), aspartate transaminase (AST), total bilirubin, Murray lung injury score, serum creatinine, eGFR, mechanical ventilation time, ICU length of stay, drug-related gastrointestinal reactions, and 30-day and 90-day all-cause mortality, among other indicators. The study aims to investigate the impact of colchicine on the levels of inflammatory factors and prognosis in patients undergoing cardiac vascular surgery and to observe the potential organ damage to the heart, lungs, liver, kidneys, and the occurrence of adverse events such as leukopenia and thrombocytopenia. This is done to assess the safety of colchicine use in cardiac surgery patients.

ELIGIBILITY:
Inclusion criteria

1. Aged between 50 and 80 years, male or female;
2. Patients undergoing elective cardiac surgery;
3. Have signed the informed consent form (ICF).

Exclusion criteria

1. Patients undergoing emergency surgery;
2. Patients undergoing deep hypothermic circulatory arrest surgery;
3. Preoperative predicted mortality >3% according to European System for Cardiac Operative Risk Evaluation II (EuroSCORE II);
4. Patients undergoing off-pump coronary artery bypass grafting (off-pump CABG) surgery;
5. Patients undergoing left or right ventricular outflow tract obstruction surgery;
6. Patients undergoing complex corrective surgery for congenital heart disease;
7. Patients with an expected CPB exceeding 180 minutes or an anticipated aortic cross-clamp time exceeding 120 minutes;
8. Patients expected to have a postoperative endotracheal tube removal time exceeding 24 hours;
9. Patients with prolonged fasting or inability to self-feed;
10. A history of malignant tumor;
11. Patients with unstable preoperative vital signs requiring intra-aortic balloon pump (IABP), extracorporeal membrane oxygenation (ECMO)assistance, or endotracheal tube-assisted ventilation;
12. A history of cardiac surgery;
13. Patients with preoperative gastrointestinal symptoms, such as nausea, vomiting and diarrhea;
14. Patients with a history of dialysis before surgery;
15. Patients with a history of atrial fibrillation before surgery;
16. Patients on long-term hepatorenal protective medications;
17. Patients with hepatic and renal insufficiency (Child-Pugh class B or C, estimated glomerular filtration rate <35 mL/min/1.73 m2);
18. Patients with abnormal baseline inflammatory markers [interleukin-6 (IL6) >10 pg/mL, procalcitonin (PCT) >0.5 ng/mL, C reactive protein (CRP) >10 mg/L];
19. Patients diagnosed with infectious diseases, inflammatory immune diseases, or tumor;
20. Patients who have received immunosuppressive or anti-inflammatory treatment;
21. Patients allergic or intolerant to colchicine;
22. Breastfeeding or pregnant women;
23. Other situations deemed inappropriate for participation in the study by the investigator.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 768 (Estimated)
Dates: Start 2024-01-28 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with POAF | postoperative 10 days
  POAF: Onset of new atrial fibrillation in patients within 10 days post-surgery.
Number of Participants with PMI | postoperative 10 days
  PMI: Patient's high-sensitivity cardiac troponin T (hs-cTnT) exceeds 0.8 ng/L on the first day after surgery, and there is an increase of 10% or more on the second day compared to the first day postoperatively.
Number of Participants with ARDS | postoperative 10 days
  ARDS: Acute Respiratory Distress Syndrome
Number of Participants with PPS | postoperative 10 days
  PPS: post-pericardiotomy syndrome

SECONDARY OUTCOMES:
Oxygenation index | postoperative day 1, 3, 5 and 7
  SpO2 /FIO2
Inflammatory index | postoperative day 1, 3, 5 and 7
  WBC[×109/L], Neutrophil[NEU,%], Interleukin(IL)-1β[pg/mL], IL-6[pg/mL], IL-8[pg/mL], TNF-α[pg/mL], CRP[mg/L], PCT[ng/mL], neutrophil elastase[NE,ng/mL] and myeloperoxidase[MPO, ng/ml]
Myocardial injury marker | postoperative day 1, 3, 5 and 7
  myoglobin[Myo, ng/ml], CK-MB[ng/ml], hs-cTnT[ng/ml]
Acute physiology and chronic health evaluation(APACHE II) socre | postoperative day 1, 3, 5 and 7
  Interpretation of APACHE II : minimum 0 and maximum 71; increasing score is associated with an increasing risk of hospital death. acute physiology score, chronic health status score, and age adjustment score
Murray lung injury score | postoperative day 1, 3, 5 and 7
  0 score - Indicates no lung injury; Less than 2.5 score - Indicates mild to moderate lung injury; More than 2.5 score - Indicates presence of severe ARDS. rs: respiratory rate, oxygenation, temperature, blood pressure, heart rate, and mental status
Liver and kidney function | postoperative day 1, 3, 5 and 7
  ALT[U/L], AST[U/L], BUN[mmol/L], creatinine[μmol/L], eGFR[mL/min/1.73m2], total bilirubin[mg/dL]
DVMV | postoperative 28 days
  Duration of mechanical ventilation
ICU time | postoperative 28 days
  Time to stay in the intensive care unit
In-hospital time | postoperative 28 days
  All time during hospitalization
30-day all-cause mortality | postoperative 30 days
  Proportion of deaths caused by various reasons within a certain period of time (30 days) compared to the total number of people in a certain group
90-day all-cause mortality | postoperative 90 days
  Proportion of deaths caused by various reasons within a certain period of time (90 days) compared to the total number of people in a certain group
Incidence of gastrointestinal reactions | postoperative 7 days
  Adverse reactions related to colchicine
Surgical data | Surgical day
  cardiopulmonary bypass time (min)
Surgical data | Surgical day
  aortic cross-clamp time (min)
blood transfusion | Surgical day
  blood transfusion volume(ml)
Rate of exudates on chest radiograph | postoperative 14 days
  Chest radiograph on postoperative days 1, 2, and 3, and chest CT within 14 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Tuo Pan, M.D, Study Director — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School; DongJin Wang, M.D, Study Chair — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School; DongJin Wang, M.D, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Dong-Jin Wang, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li X, Luo Y, Cai X, Lv Z, Kong Y, Guo Q, Zhu J, Pan T, Wang D. Anti-inflammatory effect of colchicine on organ damage during the perioperative period of cardiac surgery: a study protocol for a multicentre, randomised, double-blind, placebo-controlled clinical trial. BMJ Open. 2024 Sep 12;14(9):e084368. doi: 10.1136/bmjopen-2024-084368. PMID 39266309